CLINICAL TRIAL: NCT04755972
Title: Mucolytic Agents and Ventilator-associated Pneumonia in Patients on Invasive Mechanical Ventilation Due to Severe Acute Respiratory Syndrome Coronavirus 2
Brief Title: Mucolytics in Patients on Invasive Mechanical Ventilation Due to Severe Acute Respiratory Syndrome Coronavirus 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Hospital Center, Split (Other)
Responsible Party: Principal Investigator, Nikola Delić, MD, intensive care specialist, Clinical Hospital Center, Split
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2181-147-01/06/M.S.-20-02
Record Dates: First submitted 2021-02-06; First posted 2021-02-16 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Corona Virus Infection; Pneumonia, Ventilator-Associated
Keywords: coronavirus disease 2019; Pneumonia, Ventilator-Associated; hypertonic saline; bicarbonate; N-acetylcysteine
MeSH Terms: conditions — Coronavirus Infections; Pneumonia, Ventilator-Associated; COVID-19 | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- N-acetylcysteine (Active Comparator): Inhalation of 5 ml-s of N-acetylcysteine every 12 hours.
  Interventions: Other: Inhalation of N-acetylcysteine
- Hypertonic saline (Active Comparator): Inhalation of 5 ml-s of 5% sodium chloride every 12 hours.
  Interventions: Other: Inhalation of 5% sodium chloride
- Bicarbonate (Active Comparator): Inhalation of 5 ml-s 8.4% sodium bicarbonate every 12 hours.
  Interventions: Other: Inhalation of 8,4% sodium bicarbonate
- Control group (No Intervention): No preventive inhalation.

INTERVENTIONS:
Other: Inhalation of N-acetylcysteine — Group 1 will receive N-acetylcysteine inhalation every 12 hours from the beginning of invasive mechanical ventilation.
  Arms: N-acetylcysteine
Other: Inhalation of 5% sodium chloride — Group 2 will receive inhalation with a 5% sodium chloride solution every 12 hours from the beginning of invasive mechanical ventilation.
  Arms: Hypertonic saline
Other: Inhalation of 8,4% sodium bicarbonate — Group 3 will receive inhalation of 8.4% sodium bicarbonate every 12 hours from the beginning of invasive mechanical ventilation.
  Arms: Bicarbonate

SUMMARY:
It is planned to include patients over 18 years of age of both sexes, admitted to the Intensive Care Unit of Clinical Hospital Centre Split for respiratory insufficiency caused by severe acute respiratory syndrome coronavirus 2 in need of invasive mechanical ventilation.

The patients will be divided into four groups. Group 1 will receive N-acetylcysteine inhalation, Group 2 will receive inhalation with a 5% sodium chloride solution, and Group 3 will receive inhalation of 8.4% sodium bicarbonate, group 4 is a control group and will not routinely receive inhaled mucolytics preventively.

All inhalations will be given twice a day 12 hours apart. The first inhalation will be included within 12 hours of the patient being enrolled in the Intensive Care Unit. Patients will be randomized according to the type of inhalation they will receive, randomization will be done by all researchers through the random.org website, and the inhalation will be given by a nurse according to the agreed protocol.

RESEARCH GOALS

The aim of this study is to determine whether there is a difference in the frequency and duration of ventilator-associated pneumonia (VAP) and whether there is a difference in the number of days spent on mechanical ventilation and in mortality in these four groups of patients.

Hypothesis

Coronavirus disease 2019 patients on invasive mechanical ventilation and preventive sodium bicarbonate inhalation will have a lower incidence of ventilator-associated pneumonia and fewer days spent on invasive mechanical ventilation than patients inhaled with N-acetylcysteine, 5% saline, or patients without preventive inhalation.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with coronavirus pneumonia who need invasive mechanical ventilation.

Exclusion Criteria:

* Patients with polytrauma,
* pregnant women,
* severe hemodynamic instability,
* patients with pulmonary edema,
* less than 3 days spent in the ICU,
* patients who have microbiologically proven bacterial infection on arrival.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-29 (Actual)

PRIMARY OUTCOMES:
Difference between 4 arms regarding ventilator-associated pneumonia rate | Through study completion, an average of 6 months.
  Patients will be monitored for ventilator-associated pneumonia according to clinical criteria with a new or progressive pulmonary infiltrate on imaging plus supportive clinical findings of infection (eg, fever, secretions, leukocytosis). The diagnosis is confirmed when lower respiratory tract sampling identifies a pathogen.

SECONDARY OUTCOMES:
Number of ventilator-free days | Day 28 after ICU admission.
  Number of days from day 1 after ICU admission and start of mechanical ventilation on which a patient breathes without assistance of the ventilator if the period of unassisted breathing lasted at least 24 consecutive hours.
Mortality | Day 28 after ICU admission.
  Life status (alive or deceased) on day 28 after ICU admission.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital Centre Split, Split, Croatia

IPD SHARING:
Plan to Share IPD: Undecided